CLINICAL TRIAL: NCT07210476
Title: Turkish Adaptation and Psychometric Evaluation of the Sleep Screening Tool for Children and Adolescents With Complex Chronic Conditions
Brief Title: Turkish Adaptation of a Sleep Screening Tool for Pediatric Complex Chronic Conditions
Acronym: SCAC
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Division of Social Pediatrics, Marmara University School of Medicine, Department of Pediatrics, Marmara University
Other Study IDs: 24.06.2025-73
Record Dates: First submitted 2025-07-24; First posted 2025-10-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Conditions; Pediatric Intensive Care; Sleep Disorder (Disorder); Sleep
Keywords: sleep; sleep disorder; child; chronic disease; actigraphy
MeSH Terms: conditions — Chronic Disease; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to adapt the Sleep Screening Scale for Children and Adolescents with Complex Chronic Conditions (SCAC) into Turkish and test its reliability and validity for this population. Children and adolescents with complex chronic conditions (CCC) often have ongoing and multiple health problems. These children often face a high risk of sleep problems, but there are no screening tools in Turkish designed specifically for them.

The main goal is to confirm that the Turkish version of the SCAC is accurate and reliable. The study will also look at how common different types of sleep problems are in children with CCC, and how these problems are related to factors such as diagnosis, age, sex, and other medical conditions.

Another goal is to compare children's sleep at home with their sleep during a stay in the pediatric intensive care unit (PICU). The study will also examine how environmental factors (such as light and noise) and medical factors (such as pain, medications, and devices) affect sleep in the hospital. After discharge, sleep recovery will be followed for up to 3 months using sleep diaries and actigraphy (a wearable device that measures movement during sleep).

DETAILED DESCRIPTION:
This multi-phase, prospective observational study is designed to evaluate sleep disturbances among children with complex chronic conditions (CCCs), focusing on both the hospital period-specifically pediatric intensive care units (PICUs)-and the post-discharge transition to home. The study incorporates both subjective (questionnaire-based) and objective (actigraphy-based) assessments and integrates a family-centered, developmentally appropriate, and biopsychosocial framework.

The first phase involves the cross-cultural adaptation and psychometric validation of the "Sleep Screening Tool for Children and Adolescents with Complex Chronic Conditions (SCAC)" into Turkish. This includes forward and backward translation, expert panel review, cognitive interviews with caregivers, and a pilot study. Validity (via exploratory factor analysis using principal components analysis with varimax rotation) and internal consistency (via Cronbach's alpha) will be tested. Test-retest reliability will be evaluated by re-administering the scale one month after discharge to 50 participants.

In the second phase, children admitted to one of the largest tertiary PICU in Türkiye will be recruited. During hospitalization, sleep-wake patterns will be continuously monitored using actigraphy, while environmental factors including noise and light exposure will be recorded using calibrated sensors placed at the bedside. Nurses will assist with administering tools and maintaining logs. Additional clinical variables such as medications, nighttime interventions, pain scores, and disease severity will also be recorded. The study setting enables inclusion of a high-volume and diverse pediatric population.

Following discharge, longitudinal follow-up will be conducted using the SCAC tool and sleep diaries at four time points: Day 15, Month 1, Month 2, and Month 3. Parental consent will include approval for follow-up via telephone and SMS reminders. One nurse-researcher will conduct structured phone interviews and provide diary reminders. Post-discharge sleep recovery will be evaluated based on comparison to PICU scores and pre-hospital baseline sleep as reported by parents.

This study is the first in Türkiye, to adapt and validate a sleep screening scale specifically designed for CCC. This research not only focuses on scale development but also aims to generate scientific data that could inform environmental improvements in hospital settings.

ELIGIBILITY:
Inclusion Criteria:

Age 1 month to 18 years At least one complex chronic condition (per 2014 CCC classification) Admission to a pediatric intensive care unit (PICU) Parents willing to participate Parents literate in Turkish

Exclusion Criteria:

Parents with insufficient Turkish language proficiency to complete study materials

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 1 months-18 years with at least one complex chronic condition (defined by the 2014 CCC classification)
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Psychometric validation of the Turkish version of the Sleep Screening Scale for Children and Adolescents with Complex Chronic Conditions (SCAC) | At enrollment (hospitalization)
  Description: The primary outcome is the psychometric validation of the Sleep Screening Scale for Children and Adolescents with Complex Chronic Conditions (SCAC), originally developed by Larissa Alice Kubek and adapted into Turkish (Kronik Karmaşık Durumu Olan Çocuklar ve Ergenler İçin Uyku Tarama Anketi; KUBA) through forward-backward translation. The scale consists of 29 items grouped into four factors based on the International Classification of Sleep Disorders - Third Edition (ICSD-3) diagnostic categories:
  Sleep initiation and maintenance (7 items)
  Sleep-related breathing and arousals (9 items)
  Daytime sleepiness (7 items)
  Sleep-related movements (6 items)
  Each item is rated for the frequency of symptoms in the past 7 days, with higher scores indicating a greater presence of sleep-related problems. The total score ranges from 0 to 203, and subscale scores range from 0 to 63 depending on the number of items in each factor. Internal consistency will be assessed using Cronbach's
Test-retest reliability of the Turkish version of the SCAC | At least 4 weeks post-discharge from PICU
  Test-retest reliability will be assessed in a subgroup of participants by re-administering the SCAC at least four weeks after discharge from the pediatric intensive care unit (PICU). Reliability will be calculated using intraclass correlation coefficients (ICCs) for the total and subscale scores
Prevalence and subtype distribution of sleep disturbances in children with Complex Chronic Conditions (CCC) | At enrollment (hospitalization)
  Sleep disturbances will be assessed using the SCAC Scale. The questionnaire has 29 items; each item is rated for frequency of occurrence in the past 7 days (0 = never, 7 = every day). Four subscale scores are calculated based on the SCAC domains: (1) Sleep initiation and maintenance (7 items, score range 0-49), (2) Sleep-related breathing and arousals (9 items, score range 0-63), (3) Daytime sleepiness (7 items, score range 0-49), and (4) Sleep-related movements (6 items, score range 0-42). The total score ranges from 0 to 203, with higher scores indicating greater presence of sleep-related problems.

SECONDARY OUTCOMES:
Objective sleep parameters during PICU stay | During PICU hospitalization (up to 30 days)
  Objective sleep will be assessed using wrist actigraphy, placed on Day 1 of PICU admission in participants for whom actigraphy is feasible, and corroborated with sleep diaries and nursing observation logs. The primary reported metric will be sleep efficiency, calculated as total sleep time ÷ total sleep opportunity × 100% per night and averaged across the PICU stay. Higher percentages indicate better sleep efficiency. Additional exploratory parameters (total sleep time, number of awakenings, longest uninterrupted sleep period) will be collected to characterize sleep patterns and for quality checks, but not as separate outcome measures.
Correlation of environmental and clinical factors with sleep efficiency (actigraphy and sleep diaries) | From Day 1 of PICU admission through discharge (up to 30 days)
  The primary outcome will be sleep efficiency measured using actigraphy and daily sleep diaries. Sleep efficiency will be calculated as: total sleep time ÷ total sleep opportunity × 100%, and averaged across the PICU stay. Correlation analyses will be conducted between sleep efficiency and: Light exposure (lux; actigraphy ambient light channel), Sound exposure (dB; bedside calibrated sound level meter), Nighttime nursing interventions (nursing observation logs), Pain (Face, Legs, Activity, Cry, Consolability scale, (0-10) ; Numeric Rating Scale (0-10)) Disease severity (Pediatric Logistic Organ Dysfunction-2 daily score) Medication exposure (yes/no, for sedatives, and related medications).
  Exploratory sleep parameters will also be derived from actigraphy and diaries, including:
  Total sleep time (minutes/night), Number of awakenings (count/night), Longest uninterrupted sleep period (minutes/night). These will be reported for descriptive analyses but not as separate outcome measures
Comparison of home and hospital sleep patterns | Home baseline: parent-reported 7 days prior to admission; PICU: Day 7 of admission or at discharge if earlier
  Sleep patterns will be assessed with the SCAC in Complex chronic conditions. Parents will report the home baseline sleep over the previous 7 days before admission, and the SCAC will be administered in the PICU on Day 7 of admission or at discharge whichever comes first. The outcome will be the change in SCAC scores. SCAC total scores range from 0-203; higher scores indicate greater sleep-related problems.
Change in SCAC Scores From Hospitalization to 3 Months Post-Discharge | Baseline (hospitalization),15 days, 1,2, 3 months post-discharge
  Sleep problems will be assessed with the SCAC after discharge. SCAC will be administered at Day 15, Month 1, Month 2, and Month 3 post-discharge. The primary reported value is the change in SCAC scores from hospitalization to Month 3. SCAC total score range: 0-203; higher scores indicate worse sleep-related problems.
Time to Return to Pre-Hospital Sleep-Wake Pattern | Baseline (hospitalization),15 days, 1,2, 3 months post-discharge
  Caregiver-completed sleep diaries and wake time logs will be used to monitor bedtime, wake time, and daytime napping patterns from hospitalization through 3 months post-discharge. Pre-hospital baseline is defined as the parent-reported sleep diary for the 7 days prior to admission. "Recovery" will be defined as the first date on which the sleep-wake schedule returns to the caregiver's perception of the child's typical pre-hospital pattern, based on diary entries. The primary reported value is the number of days from hospital discharge to recovery (censored at 90 days)
Correlation of clinical and environmental factors with delayed recovery of sleep-wake patterns | From hospital discharge through 90 days post-discharge
  Delayed recovery is defined as return to the baseline sleep-wake pattern (caregiver-completed sleep diaries) occurring later than the median recovery time in the study cohort. The primary reported value will be time to recovery (days) after hospital discharge.
  Correlation analyses will be conducted with the following predictors:
  Disease severity: Pediatric Logistic Organ Dysfunction-2 (PELOD-2) daily score,
  Complex Chronic Condition (CCC) subtype: e.g., neurologic, cardiac, metabolic, other,
  ICU length of stay: days,
  Baseline sleep problems: SCAC total score (0-203),
  Environmental stressors:
  Light exposure (lux; measured by actigraphy ambient light channel),
  Sound exposure (dB; bedside calibrated sound level meter).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Department of Pediatrics, Division of Social Pediatrics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon reasonable request depending on ethical approvals, participant consent, and institutional policies. Any data sharing will follow strict guidelines to ensure confidentiality and data protection, especially due to the involvement of pediatric patients with complex medical conditions. Requests for sharing of individual participant data will be evaluated on a case-by-case basis. If researchers express interest (e.g., based on publications or institutional announcements), data sharing requests can be submitted through a formal application process.
Supporting Information: Study Protocol
Time Frame: Available after study completion and publication, for at least 3 years
Access Criteria: Researchers with methodologically sound proposals may request access by contacting the corresponding author. Data will be shared in accordance with ethical approval and institutional policies.

REFERENCES:
- [Background] Kubek LA, Claus B, Rostasy K, Bertolini A, Schimmel M, Fruhwald MC, Classen G, Zernikow B, Wager J. Development and preliminary validation of the Sleep Screening for Children and Adolescents with Complex Chronic Conditions (SCAC). J Sleep Res. 2023 Aug;32(4):e13881. doi: 10.1111/jsr.13881. Epub 2023 Mar 16. PMID 36929532
- [Background] Comrey AL. Factor-analytic methods of scale development in personality and clinical psychology. J Consult Clin Psychol. 1988 Oct;56(5):754-61. doi: 10.1037//0022-006x.56.5.754. No abstract available. PMID 3057010
- [Background] Kudchadkar SR, Aljohani OA, Punjabi NM. Sleep of critically ill children in the pediatric intensive care unit: a systematic review. Sleep Med Rev. 2014 Apr;18(2):103-10. doi: 10.1016/j.smrv.2013.02.002. Epub 2013 May 21. PMID 23702219
- [Background] Knauert MP, Ayas NT, Bosma KJ, Drouot X, Heavner MS, Owens RL, Watson PL, Wilcox ME, Anderson BJ, Cordoza ML, Devlin JW, Elliott R, Gehlbach BK, Girard TD, Kamdar BB, Korwin AS, Lusczek ER, Parthasarathy S, Spies C, Sunderram J, Telias I, Weinhouse GL, Zee PC. Causes, Consequences, and Treatments of Sleep and Circadian Disruption in the ICU: An Official American Thoracic Society Research Statement. Am J Respir Crit Care Med. 2023 Apr 1;207(7):e49-e68. doi: 10.1164/rccm.202301-0184ST. PMID 36999950
- [Background] Hybschmann J, Topperzer MK, Gjaerde LK, Born P, Mathiasen R, Sehested AM, Jennum PJ, Sorensen JL. Sleep in hospitalized children and adolescents: A scoping review. Sleep Med Rev. 2021 Oct;59:101496. doi: 10.1016/j.smrv.2021.101496. Epub 2021 Apr 26. PMID 33984632
- [Background] Berger J, Zaidi M, Halferty I, Kudchadkar SR. Sleep in the Hospitalized Child: A Contemporary Review. Chest. 2021 Sep;160(3):1064-1074. doi: 10.1016/j.chest.2021.04.024. Epub 2021 Apr 22. PMID 33895129
- [Background] Adavadkar PA, Brooks L, Pappalardo AA, Schwartz A, Rasinski K, Martin MA. Association between sleep disorders and health care utilization in children with chronic medical conditions: a Medicaid claims data analysis. J Clin Sleep Med. 2024 Apr 1;20(4):595-601. doi: 10.5664/jcsm.10936. PMID 38217477
- [Background] Namisango E, Bristowe K, Allsop MJ, Murtagh FEM, Abas M, Higginson IJ, Downing J, Harding R. Symptoms and Concerns Among Children and Young People with Life-Limiting and Life-Threatening Conditions: A Systematic Review Highlighting Meaningful Health Outcomes. Patient. 2019 Feb;12(1):15-55. doi: 10.1007/s40271-018-0333-5. PMID 30361884
- [Background] Dreier LA, Zernikow B, Stening K, Wager J. Insights into the Frequency and Distinguishing Features of Sleep Disorders in Pediatric Palliative Care Incorporating a Systematic Sleep Protocol. Children (Basel). 2021 Jan 17;8(1):54. doi: 10.3390/children8010054. PMID 33477321
- [Background] Shelton AR, Malow B. Neurodevelopmental Disorders Commonly Presenting with Sleep Disturbances. Neurotherapeutics. 2021 Jan;18(1):156-169. doi: 10.1007/s13311-020-00982-8. Epub 2021 Jan 5. PMID 33403472
- [Background] Blackmer AB, Feinstein JA. Management of Sleep Disorders in Children With Neurodevelopmental Disorders: A Review. Pharmacotherapy. 2016 Jan;36(1):84-98. doi: 10.1002/phar.1686. PMID 26799351
- [Background] Bai G, Herten MH, Landgraf JM, Korfage IJ, Raat H. Childhood chronic conditions and health-related quality of life: Findings from a large population-based study. PLoS One. 2017 Jun 2;12(6):e0178539. doi: 10.1371/journal.pone.0178539. eCollection 2017. PMID 28575026
- [Background] Xavier WDS, Abreu MP, Nunes MDR, Silva-Rodrigues FM, da Silva LF, de Araujo BBM, De Bortoli PS, Neris RR, Nascimento LC. The Sleep Patterns of Children and Adolescents with Chronic Conditions and Their Families: An Integrative Literature Review. Children (Basel). 2024 Feb 6;11(2):207. doi: 10.3390/children11020207. PMID 38397320
- [Background] Feudtner C, Feinstein JA, Zhong W, Hall M, Dai D. Pediatric complex chronic conditions classification system version 2: updated for ICD-10 and complex medical technology dependence and transplantation. BMC Pediatr. 2014 Aug 8;14:199. doi: 10.1186/1471-2431-14-199. PMID 25102958
- [Background] Oliveira PV, Enes CC, Nucci LB. How are children with medical complexity being identified in epidemiological studies? A systematic review. World J Pediatr. 2023 Oct;19(10):928-938. doi: 10.1007/s12519-022-00672-9. Epub 2022 Dec 27. PMID 36574212
- [Background] Marcus KL, Kao PC, Ma C, Wolfe J, DeCourcey DD. Symptoms and Suffering at End of Life for Children With Complex Chronic Conditions. J Pain Symptom Manage. 2022 Jan;63(1):88-97. doi: 10.1016/j.jpainsymman.2021.07.010. Epub 2021 Jul 24. PMID 34311060